CLINICAL TRIAL: NCT05791461
Title: Stress in Working Life - Realist Evaluation of a Stress Management Intervention for Patients Referred to an Occupational Health Clinic Due to Work-related Stress
Brief Title: Stress in Working Life
Status: Recruiting | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IOB_SDU_CBB_LNA
Record Dates: First submitted 2023-02-23; First posted 2023-03-30 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Occupational Stress
Keywords: Occupational stress; Cognitive behavioural therapy; Realist evaluation
MeSH Terms: conditions — Occupational Stress | interventions — Mars

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention cohort: Patients with work-related stress (F43.2/8/9 or Z56.3 (ICD-0)) who received the stress management intervention between 2011-2018 (N>400). The intervention is based on cognitive behavioral therapy, delivered by a trained psychologist in groups of 8-10 patients. The intervention consists of 8 sessions in 3 months, with a booster session 3 months after the intervention has ended.
  Interventions: Behavioral: MARS (Measures Against Work-related Stress)
- Comparison cohort: Patients with work-related stress (diagnoses F43.2/8/9 or Z56.3 (ICD-10)) who was seen at a consultation at Department of Occupational and Environmental Health in Odense (DOEM) in 2011-2012, but did not receive the intervention because it was not yet offered. The patients were offered advice and support by a psychologist (usual care). The intervention was introduced at DOEM in 2011 for a limited number of patients due to introducing the intervention and establishing the capacity of psychologists involved. In 2013 the intervention was implemented at full scale to include every eligible patient.

INTERVENTIONS:
Behavioral: MARS (Measures Against Work-related Stress) — The stress management intervention is based on cognitive behavioral therapy and aims to change the way patients perceive and cope with stressful situations at work.
  It is group sessions over 3 months with approximately 9 participants. Participants meet 9 times (once a week the first 3 weeks and once every second week the last 5 times) and for a follow-up session 3 months after the intervention has ended. Each session lasts for 3 hours and is led by a trained psychologist. The participants perform tasks at home between the sessions. In the first session the rationale behind the intervention is introduced. In session 2 and 3 the patients work with enhancing self-regulation. In session 4 and 5 the focus is on modifying intermediate beliefs. In session 6 the focus is on improving interaction. Session 7 and 8 focuses on consolidation of learning and strategies to prevent relapse, and session 9 is a follow-up session 3 months after the intervention has ended.
  Groups: Intervention cohort

SUMMARY:
The goal of this realist evaluation of a Danish Cognitive Behavioral Therapy (CBT)-based stress management for patients with work-related stress is to understand what works, for whom, in what circumstances.The main objectives are:

To assess the effect of the stress management intervention on sustainable return to work.

To investigate what contexts and mechanisms are associated with patients' return to work rates and level of perceived stress after having received the stress management intervention.

To understand from a patient perspective how mechanisms work in specific contexts to generate effects of the stress management intervention.

The evaluation comprises two observational studies and one interview study. The intervention cohort are patients with work-related stress who received the stress management intervention between 2012-2018.

The comparison cohort are patients who would have been eligible to receive the intervention in 2011-2012, however they did not receive any intervention because it was not offered at that time.

In study one return to work rates are compared between the intervention cohort and the comparison cohort to find out if the intervention can help patients return to work at a faster rate.

Study two will investigate if there are any explanatory variables (such as work type, civil status or level of depressive symptoms) that may explain why some patients benefit more or less from the intervention.

Study three will explore what it is about the intervention (mechanisms) the patients find are helping them to cope with stress or the opposite in specific circumstances.

ELIGIBILITY:
Inclusion Criteria:

* exposure to stressful conditions at work such as a large workload and/or stressful organisational and managerial conditions.
* Patients must be employed, and if on sick leave there must be plans for return to work during the intervention period.
* Patients must exhibit severe signs of work-related stress meaning that there must have been a significant work-related impact, the patient must have had physical, psychological, and behavioural stress symptoms for more than four weeks.

Exclusion Criteria:

* patient's work-related stress is primarily caused by cooperation problems, bullying and/or harassment,
* long-term sick leave >26 weeks up to referral
* more severe stress load outside of work
* severe psychiatric conditions that requires treatment
* current abuse of alcohol and/or psychoactive stimulants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with work-related stress (diagnoses F43.2/8/9 or Z56.3 (ICD-10)) seen at Department of Occupational and Environmental Medicine, Odense, in the period 2011-2018
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The effect of the stress management intervention on sustainable return to work (RTW). | 36 months after first contact with clinic.
  The primary outcome is sustainable RTW which is defined as returning to full-time work for a minimum of four months without any sick-leave compensation. Data from the DREAM database (national database containing information about sick leave compensation in the Danish population) will be obtained for both the intervention cohort and the comparison cohort for the two-year period prior to the first consultation at Department of Occupational and Environmental Medicine, Odense, and for three years after.
Identification of possible contexts and mechanisms associated with patients' RTW rates after having received the stress management intervention. | 36 months after first contact with clinic.
  Data on sick leave compensation from the DREAM database.
From a patient perspective how mechanisms work in specific contexts to generate effects of the stress management intervention. | Up to 12 months after intervention.
  From realist theory driven interviews patient-reported context-mechanism -outcome-configurations will be used to refine, confirm or refute the initial program theory.

CONTACTS AND LOCATIONS:
Overall Officials: Lotte N Andersen, PhD, Study Chair — University of Southern Denmark
Locations (1):
- Department of Occupational and Environmental Medicine, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No